CLINICAL TRIAL: NCT06691958
Title: Impact of Chip Thickness and Size on Eating Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2409
Record Dates: First submitted 2024-11-11; First posted 2024-11-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-05

CONDITIONS: Consumer Behavior; Consumer Preference; Consumer Satisfaction
Keywords: sensory testing; intake; calories; duration of eating; rate of consumption; snack; liking; satiation; chewing; emotion; satisfaction; fullness
MeSH Terms: conditions — Consumer Behavior; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Standard tortilla chip for Sensory Study (Active Comparator): Snack comparable to marketed version
  Interventions: Other: Tortilla corn chips 4-5 pieces, eat one piece at time
- Thicker than standard tortilla chip with same amount of seasoning per 100g for Sensory Study (Experimental): Snack
  Interventions: Other: Tortilla corn chips 4-5 pieces, eat one piece at time
- Standard extruded chip for Sensory Study (Active Comparator): Snack comparable to marketed version
  Interventions: Other: Extruded corn chips 4-5 pieces, eat one piece at time
- Bigger extruded chip with same seasoning per 100g for Sensory Study (Experimental): Snack
  Interventions: Other: Extruded corn chips 4-5 pieces, eat one piece at time
- Bigger extruded chip with same concentration of seasoning on surface per 100g for Sensory Study (Experimental): Snack
  Interventions: Other: Extruded corn chips 4-5 pieces, eat one piece at time
- Standard tortilla chip for Ad libitum Study (Active Comparator): Snack comparable to marketed version
  Interventions: Other: Tortilla corn chips 90 grams
- Thicker than standard tortilla chip with same seasoning per 100g for Ad libitum Study (Experimental): Snack
  Interventions: Other: Tortilla corn chips 90 grams
- Standard extruded chip for Ad libitum Study (Active Comparator): Snack comparable to marketed version
  Interventions: Other: Extruded corn chips 90 grams
- Bigger extruded chip with same seasoning per 100g for Ad libitum Study (Experimental): Snack
  Interventions: Other: Extruded corn chips 90 grams
- Bigger extruded chip with same concentration of seasoning on surface per 100g for Ad libitum Study (Experimental): Snack
  Interventions: Other: Extruded corn chips 90 grams

INTERVENTIONS:
Other: Tortilla corn chips 4-5 pieces, eat one piece at time — Snack
  Arms: Standard tortilla chip for Sensory Study; Thicker than standard tortilla chip with same amount of seasoning per 100g for Sensory Study
Other: Tortilla corn chips 90 grams — Snack
  Arms: Standard tortilla chip for Ad libitum Study; Thicker than standard tortilla chip with same seasoning per 100g for Ad libitum Study
Other: Extruded corn chips 90 grams — Snack
  Arms: Bigger extruded chip with same concentration of seasoning on surface per 100g for Ad libitum Study; Bigger extruded chip with same seasoning per 100g for Ad libitum Study; Standard extruded chip for Ad libitum Study
Other: Extruded corn chips 4-5 pieces, eat one piece at time — Snack
  Arms: Bigger extruded chip with same concentration of seasoning on surface per 100g for Sensory Study; Bigger extruded chip with same seasoning per 100g for Sensory Study; Standard extruded chip for Sensory Study

SUMMARY:
To analyze prototypes developed with the base and seasonings of products that exhibit variations in chip thickness and size. The information obtained from this analysis will serve as the basis for subsequent research to explore different prototype options with increased satiation properties.

DETAILED DESCRIPTION:
There are two study components, a sensory study and an ad libitum study. Eighty-eight participants will test tortilla chips and eighty-eight will test extruded chips in the sensory study. On a first-come first-served basis, forty-four of the eighty-eight chip participants from the sensory testing phase will test tortilla chips, and forty-four of the eighty-eight extruded chip participants will test extruded chips in the ad libitum study.

ELIGIBILITY:
Inclusion Criteria:

* Report eating tortilla and/or extruded chips regularly, non-rejector of cheese flavor chips
* Provide informed consent
* Speak and understand English without difficulty
* Willing to eat similar food the day prior and on the day of each visit to the testing facility for ad libitum sessions
* Describe yourself as generally healthy

Exclusion Criteria:

* Those who are on restricted diet due to a weight loss or maintenance purpose
* Participants with class III occlusions for ad libitum sessions
* Have abnormal taste, chewing and smell ability
* Smoke or vape
* Being pregnant or breastfeeding
* Allergic or intolerance to any of the product ingredients (section 6), especially milk and wheat
* Participation in a sensory clinical trial within past 7 days (we do not expect carryover issue from the taste testing)
* Participation in any PepsiCo trial within past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Satiation: Intake in grams | Total grams consumed at each 30-minute ad libitum testing session from beginning of eating until end of eating on separate days, two test visits for tortilla chips arm and three test visits for extruded chips arm.
  gram weight of consumption
Satiation: Nutrition | Total calories consumed at each 30-minute ad libitum testing session from beginning of eating until end of eating on separate days, two test visits for tortilla chips arm and three test visits for extruded chips arm.
  Intake in calories
Duration of eating | Timed from beginning of eating until end of eating at each 30-minute ad libitum testing sessions on separate days, two test visits for tortilla chips arm and three test visits for extruded chips arm.
  In minutes
Rate of consumption | Measured in grams per minute at each 30-minute ad libitum testing session from beginning of eating until end of eating, on separate days, two test visits for tortilla chips arm and three test visits for extruded chips arm.
  Speed of eating in minutes
Consumer response: Liking | At end of eating each product at the one 45-minute sensory session, and at end of each 30-minute ad libitum session on separate days, two visits for the tortilla chips arm and three visits for the extruded chips arm. Higher score is the better outcome.
  9-point hedonic scale from extremely dislike to extremely like
Consumer response: Satisfaction | At end of eating each product at the one 45-minute sensory session and at end of each ad libitum session on separate days, two visits for tortilla chips arm and three visits for the extruded chips arm. Higher satisfaction is a better outcome.
  9-point hedonic scale from extremely dissatisfied to extremely satisfied
Perceived sensory properties (TCATA) | Over a period of 60 seconds for each product at the one 45-minute sensory session and at each ad libitum session on separate days, two visits for tortilla chips arm and three visits for the extruded chips arm.
  Using Temporal CATA (TCATA) choose all that apply from list of crunchy, hard, tooth clogging, loose particles, soft, airy melting
Perceived sensory properties (CATA) | Check all that apply for each product while sampling them at the one 45-minute sensory session. A favorable rating would be a better outcome.
  CATA
Emotional responses using CATA | Check all that apply for each product while sampling them at the one 45-minute sensory session. Positive ratings would be a better outcome than negative..
  Essence 25 using CATA
Hunger and Fullness and how much could you eat right now | Before eating and right after eating as much as they want to eat at each 30-minute ad libitum session on separate days, two visits for tortilla chips arm and three visits for the extruded chips arm.
  Using a 3 item Visual Analog Scale (VAS) to mark along 100 mm line the level of hunger and fullness from not at all to totally full

CONTACTS AND LOCATIONS:
Overall Officials: Qian Yang, PhD, Principal Investigator — University of Nottingham, Sensory Science Centre
Locations (1):
- University of Nottingham Sensory Science Centre, Sutton Bonington, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No